CLINICAL TRIAL: NCT00169234
Title: Immunogenicity and Safety of Varying Doses of a 7-valent Conjugate Pneumococcal Vaccine in Adults 70-79 Years of Age Who Were Previously Vaccinated With the 23-valent Pneumococcal Polysaccharide Vaccine
Brief Title: Pneumococcal Adult-dose Ranging Immunization Study
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Kaiser Permanente (Other)
Collaborators: Centers for Disease Control and Prevention (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Other
Other Study IDs: CDC Protocol 3848; CDC Task Order 0957-045 (Other Grant/Funding Number: Centers for Disease Control)
Record Dates: First submitted 2005-09-09; First posted 2005-09-15 (Estimated); Last update posted 2017-10-13 (Actual); Status verified 2017-10

CONDITIONS: Pneumonia
Keywords: Pneumococcal disease; Vaccination; Immunization; PPV23; PCV7
MeSH Terms: conditions — Pneumonia; Pneumococcal Infections | interventions — Heptavalent Pneumococcal Conjugate Vaccine; 23-valent pneumococcal capsular polysaccharide vaccine

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- 0.1mL Pneumococcal Conjugate Vaccine (Experimental): Participants in this group were randomized at enrollment to receive 0.1mL PCV7, Prevnar® at the enrollment visit and then 0.1mL Pneumococcal Polysaccharide Vaccine 12 months later.
  Interventions: Biological: PCV7, Prevnar®; Biological: Pneumovax 23
- 0.5mL Pneumococcal Conjugate Vaccine (Experimental): Participants in this group were randomized at enrollment to receive 0.5mL PCV7, Prevnar® at the enrollment visit and then 0.1mL Pneumococcal Polysaccharide Vaccine 12 months later.
  Interventions: Biological: PCV7, Prevnar®; Biological: Pneumovax 23
- 1.0mL Pneumococcal Conjugate Vaccine (Experimental): Participants in this group were randomized at enrollment to receive 1.0mL PCV7, Prevnar® at the enrollment visit and then 0.1mL Pneumococcal Polysaccharide Vaccine 12 months later.
  Interventions: Biological: PCV7, Prevnar®; Biological: Pneumovax 23
- 2.0mL Pneumococcal Conjugate Vaccine (Experimental): Participants in this group were randomized at enrollment to receive 2.0mL PCV7, Prevnar® at the enrollment visit and then 0.1mL Pneumococcal Polysaccharide Vaccine 12 months later.
  Interventions: Biological: PCV7, Prevnar®; Biological: Pneumovax 23
- 0.5mL Pneumococcal Polysacc Vaccine (Experimental): Participants in this group were randomized at enrollment to receive 0.5mL Pneumovax 23 at the enrollment visit and then 0.1mL Pneumococcal Polysaccharide Vaccine 12 months later.
  Interventions: Biological: Pneumovax 23

INTERVENTIONS:
Biological: PCV7, Prevnar® — Randomized to receive 0.1mL, 0.5mL, 1.0mL or 2.0mL at the enrollment visit, followed by 0.1mL PPV23 12 months later.
  Arms: 0.1mL Pneumococcal Conjugate Vaccine; 0.5mL Pneumococcal Conjugate Vaccine; 1.0mL Pneumococcal Conjugate Vaccine; 2.0mL Pneumococcal Conjugate Vaccine
Biological: Pneumovax 23 — Randomized to receive 0.5mL at the enrollment visit, followed by 0.1mL PPV23 12 months later.

SUMMARY:
The purpose of this study is to give seniors different doses of a new pneumococcal vaccine called PCV7 to evaluate the safety of the vaccine and compare the immune response to find out which amount gives the best immune response. The PCV7 vaccine is currently licensed by the FDA for use in infants and toddlers only.

DETAILED DESCRIPTION:
The purpose of this prospective randomized study is to assess the safety, post-vaccination antibody response, and memory response to a subsequent polysaccharide challenge of varying doses of PCV7 compared with the standard dose of PPV23 in immunocompetent adults 70-79 years of age who were previously vaccinated with PPV23 at age 65 years or above and at least 5 years previously. The study will be conducted among a total of 220 persons recruited from GHC and the Seattle VAMC. Participants will be randomized into one of 5 study groups with 44 participants per group. The antigen content of PCV7 will be varied by administration of different volumes of the licensed pediatric formulation of that vaccine. Four groups will receive one of four volumes (0.1 mL, 0.5 mL, 1.0 mL, 2.0 mL) of the licensed pediatric formulation of PCV7 followed 12 months later by administration of a challenge 0.1 mL dose of PPV23 to assess the induction of immunologic memory. The comparison group will receive the standard 0.5 mL dose of PPV23 following 12 months later by administration of a 0.1 mL dose of PPV23.

ELIGIBILITY:
Inclusion Criteria:

* Age 70 through 79 years (up to the day prior to the 80th birthday)
* Previously received exactly one dose of PPV23, and that dose was received on or after their 65th birthday and at least 5 years before the date of study enrollment
* Expected to reside in the area for at least 13 months
* Able to understand and give informed consent
* Able to perform study procedures
* Able to be contacted by telephone for follow-up on adverse events

Exclusion Criteria:

* Received >=2 doses of PPV23 prior to study enrollment.
* Living non-independently in an institutional setting, such as a nursing home. Persons living independently in adult residence communities will be eligible.
* Use of any investigational vaccine within the past 30 days or planned use during the study period.
* Current or planned participation in a research study of an investigational drug. Participation in research studies that involve use of licensed drugs, for either approved or investigational indications, will be permitted with the approval of the site PI, as will participation in research studies that do not involve medications.
* Current use or previous chronic administration, defined as >=14 days during the previous six months, of immunosuppressants or other immune-modifying drugs. (For oral or injected corticosteroids, the immune-modifying dose is defined as prednisone or its equivalent >=10 mg/day). Topical steroids are allowed.
* Current use of high doses of inhaled steroids, defined as per Table 3.
* Use of cytotoxic therapy in the previous 5 years.
* Plans to receive cytotoxic therapy during the study period.
* Receipt of parenteral immunoglobulin or blood products within three months of study.
* Plans to receive parenteral immunoglobulin or blood products within the study period.
* Current ongoing use of warfarin or heparin or has a bleeding disorder, such as ITP.
* Any confirmed or suspected immunosuppressive or immunodeficient condition, including human immunodeficiency virus (HIV) infection.
* Anatomic or known functional asplenia.
* History of a hematologic malignancy or a pre-malignant condition (i.e., leukemia, lymphoma, multiple myeloma, myelodysplasia).
* Active neoplastic disease, excluding local skin cancer or other malignancies (e.g. prostate cancer) that are stable in the absence of immunosuppressive/cytotoxic or radiation therapy.
* End-stage liver disease or hepatic failure (as diagnosed by a physician or evidenced by a history within the last 10 years of bleeding esophageal varices, ascites, or hepatic encephalopathy).
* Renal failure, as evidenced by current or expected dialysis or known creatinine of >=2.5 ug/ml.
* Known hypersensitivity to PPV23 or to any component of PPV23 or PCV7, including aluminum phosphate or diphtheria protein.
* Presence of any other condition or impairment that in the opinion of the investigator is likely to compromise the participant's ability to complete the study procedures.

Ages: 70 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 220 (Actual)
Dates: Start 2003-05; Primary Completion 2005-02 (Actual); Study Completion 2005-02 (Actual)

PRIMARY OUTCOMES:
To evaluate the immunologic response to varying doses of 7-valent pneumococcal conjugate vaccine (PCV7) among older adults. | Pre/post enrollment vaccination, and pre/post 1 year challenge vaccination

SECONDARY OUTCOMES:
To evaluate the safety to varying doses of 7-valent pneumococcal conjugate vaccine (PCV7) among older adults. | During the 13 month study period.

CONTACTS AND LOCATIONS:
Overall Officials: Lisa A Jackson, MD, MPH, Principal Investigator — Kaiser Permanente
Locations (2):
- United States (2):
  - Group Health Research Institute, Seattle, Washington
  - VA Puget Sound Health Care System, Seattle, Washington

REFERENCES:
- [Result] Jackson LA, Neuzil KM, Nahm MH, Whitney CG, Yu O, Nelson JC, Starkovich PT, Dunstan M, Carste B, Shay DK, Baggs J, Carlone GM. Immunogenicity of varying dosages of 7-valent pneumococcal polysaccharide-protein conjugate vaccine in seniors previously vaccinated with 23-valent pneumococcal polysaccharide vaccine. Vaccine. 2007 May 16;25(20):4029-37. doi: 10.1016/j.vaccine.2007.02.062. Epub 2007 Mar 12. PMID 17391816
- [Result] Jackson LA, Neuzil KM, Whitney CG, Starkovich P, Dunstan M, Yu O, Nelson JC, Feikin DR, Shay DK, Baggs J, Carste B, Nahm MH, Carlone G. Safety of varying dosages of 7-valent pneumococcal protein conjugate vaccine in seniors previously vaccinated with 23-valent pneumococcal polysaccharide vaccine. Vaccine. 2005 May 25;23(28):3697-703. doi: 10.1016/j.vaccine.2005.02.017. PMID 15882530